CLINICAL TRIAL: NCT06407336
Title: Comparative Effect of Cylindrical Lenses Verses Spherical Equilient on Contrast Sensitivity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/702
Record Dates: First submitted 2024-05-02; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Low Vision Aids
MeSH Terms: interventions — Contrast Sensitivity; Refraction, Ocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contrast sensitivity (Experimental)
  Interventions: Diagnostic Test: Contrast sensitivity
- Refraction (Other)
  Interventions: Other: Refraction

INTERVENTIONS:
Diagnostic Test: Contrast sensitivity — Contrast sensitivity will be assessed by using two different techniques of refraction on is Cylinderical lens and other is Spherical equivalent
  Arms: Contrast sensitivity
Other: Refraction — Refraction will be performed and contrast sensitivity will be assessed to assess patient comfort level and compliance.
  Arms: Refraction

SUMMARY:
the concept of spherical equivalent plays a pivotal role in simplifying the prescription and enhancing communication between eye care professionals and patients. The spherical equivalent is a calculated value that condenses the spherical and cylindrical components into a single power.

DETAILED DESCRIPTION:
Mathematically, it is determined by adding half of the cylindrical power to the spherical power (SE = Sphere + (Cylinder/2)). This calculated value serves as a convenient representation of the overall refractive error, aiding in a more straightforward understanding of the prescription. Understanding their individual and collective impact on contrast sensitivity opens up new avenues for refining corrective interventions and enhancing the overall quality of vision. This article aims to demystify the intricate relationship between spherical equivalent and cylindrical correction, and their collective impact on contrast sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 18 to 35 years will be included.
* Both genders will be included.
* Patients having astigmatism will be included.
* Patients having 6/6 corrected vision will be included.
* Eyes having no other ocular pathology will be included.
* Patients having no history of ocular surgery or corneal scar will be included.

Exclusion Criteria:

* i. Eyes having any ocular pathology will be excluded.
* Patients with corneal suture will be excluded.
* Those using contact lenses instead of spectacles for vision correction will be excluded.
* Participants with a history of eye surgery within the past year will be excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Contrast sensitivity | 12 Months
  The ability to perceive sharp and clear outlines of very small objects. It is also defined as the ability to identify minute differences in the shadings and patterns. CS helps detect objects without a clear outline and distinguish them from their background contrast

CONTACTS AND LOCATIONS:
Locations (1):
- Sehat Medical Complex Hanjarwal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No